CLINICAL TRIAL: NCT00032552
Title: CSP #476DP - Enhancing Quality of Informed Consent (EQUIC-DP) Developmental Phase
Brief Title: Enhancing Quality of Informed Consent (EQUIC-DP) Developmental Phase
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Lavori, Philip - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: 476DP
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Informed Consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Patients in 'parent' cooperative studies projects are interviewed about their experiences in the informed consent process.

DETAILED DESCRIPTION:
Intervention: Immediately after giving informed consent for the parent study and before randomization, research subjects will be asked for consent to participate in EQUIC-DP.

The parent-study staff will provide the research subject with privacy and place a call to the coordinating center. Staff (at the EQUIC coordinating center), who will be administering the Brief Informed Consent Evaluation Protocol (BICEP) to the research subject, will introduce themselves. Then, the subject will be interviewed using a BICEP structured assessment questionnaire of approximately 12-20 open ended questions, aimed at determining the success and validity of the informed consent process of the parent study. The results of the interviews will be used to fine-tune and adjust both the process of assessing informed consent in this manner as well as the questionnaire itself.

Primary Hypothesis: Enhancing the Quality of Informed Consent Development Phase (EQUIC-DP) is a pilot and instrument-development study that will be used as the base for a VA Cooperative Studies Program-wide initiative on informed consent, called EQUIC (Enhancing the Quality of Informed Consent). EQUIC-DP has as its primary aim the field testing and iterative improvement of a method for measuring the success of an informed consent encounter with a patient-subject.

Primary Outcomes: The quality of the informed consent process, as measured by the BICEP (Brief Informed Consent Evaluation Protocol). The BICEP also offers a method to certify informed consent in routine use.

Study Abstract: Practitioners of clinical trials have a responsibility to ensure that patients participation in research is informed and voluntary. This implies that we should continuously strive to improve the effectiveness of methods for informing prospective research volunteers about experimental studies, thereby enhancing the likelihood that their interests are respected. Innovations in informed consent should be tested in realistic contexts (i.e., in clinical trials) and when appropriate with randomization at the first opportunity. In this proposed project we take efforts to improve the quality of informed consent, based on experimentation with informed consent in ongoing clinical trials in the VA Cooperative Studies Program. The CSP is uniquely situated to serve as a testing ground for informed consent, not only because of concerns for enhancing consent for human experimentation, but also because of the centralized coordination of wide variety of clinical studies representing an extraordinary range of patient capacities and vulnerabilities. Moreover, such an effort is a special responsibility of the VA given the profound trust placed in the research enterprise by veterans.

ELIGIBILITY:
Inclusion Criteria:

Depends on 'parent' study

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Veterans
Sampling Method: Non-Probability Sample
Enrollment: 632 (Actual)
Dates: Start 1999-04; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
measuring the process and outcome if informed consent | immediately during patient interview

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lavori, PhD, Study Chair — VA Palo Alto Health Care System
Locations (18):
- United States (18):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - VA Palo Alto Health Care System, Palo Alto, California
  - MIMA Century Research Assoc. (CSP #424) (DP), Melbourne, Florida
  - West Palm Beach VA Medical Center, West Palm Beach, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Rochester (CSP #424) (DP), Rochester, Minnesota
  - VA Medical Center, St Louis, St Louis, Missouri
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Northport, Northport, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington